CLINICAL TRIAL: NCT02658812
Title: A Phase II Study Using Talimogene Laherparepvec for Inflammatory Breast Cancer (IBC) or Non-IBC Patients With Inoperable Local Recurrence
Brief Title: Talimogene Laherparepvec in Treating Patients With Recurrent Breast Cancer That Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Per PI
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0034; NCI-2016-00199 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0034 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2016-01-14; First posted 2016-01-20 (Estimated); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Malignant Chest Wall Neoplasm; Recurrent Breast Carcinoma; Recurrent Inflammatory Breast Carcinoma; Stage IV Breast Cancer AJCC v6 and v7; Stage IV Inflammatory Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (talimogene laherparepvec) (Experimental): Patients receive talimogene laherparepvec IT on day 1. Cycles repeat every 3 weeks in cycle 1 and every 2 weeks thereafter in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Talimogene Laherparepvec

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Talimogene Laherparepvec — Given IT
  Other Names: ICP34.5-, ICP47-deleted Herpes Simplex Virus 1 (HSV-1) Incorporating the Human GM-CSF Gene; Imlygic; JS1 34.5-hGMCSF 47- pA-; T-VEC

SUMMARY:
This phase II trial studies how well talimogene laherparepvec works in treating patients with breast cancer that has come back and cannot be removed by surgery. Biological therapies, such as talimogene laherparepvec, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop cancer cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of talimogene laherparepvec in inflammatory breast cancer or non-inflammatory breast cancer patients with inoperable local recurrence measured by the overall response rate.

SECONDARY OBJECTIVES:

I. To determine the efficacy of talimogene laherparepvec in inflammatory breast cancer or non-inflammatory breast cancer patients with inoperable local recurrence measured by the overall disease control rate.

II. To determine the rate of local overall response and disease control rate, progression-free survival (PFS), and overall survival (OS) in all patients.

III. To determine the rate of local overall response and disease control rate, PFS, and OS in patients without distant metastases.

IV. To determine the rate of local overall response and disease control rate, PFS, and OS in patients with distant metastases.

V. To determine the safety of talimogene laherparepvec injection to local disease.

CORRELATIVE STUDIES:

I. To determine the effect of talimogene laherparepvec on injection sites and distant metastatic sites by evaluating immune function and apoptosis with immune cell surface markers and cytokines.

II. To assess changes in the following: serum or plasma levels of interleukin (IL)-2, IL-12, tumor necrosis factor (TNF)-alpha, and interferon (IFN)- alpha; (Reuben's Lab); phenotype for T-cell subsets (CD3, CD4, CD8, CD25) and natural killer cell (NK-cell) subsets (CD16, CD56), which will be determined via multiparameter fluorescence-activated cell sorting (FACS) analysis (percentage and absolute numbers) in peripheral blood at Dr. James Reuben's laboratory of MD Anderson; serum analysis of herpes simplex virus (HSV) type 1 serology with immunoglobulin (Ig)G and IgM (enzyme-linked immunosorbent assay [ELISA]).

III. To assess distant tumor tissue changes by evaluating necrosis and immune cell infiltration (T-/B-/NK-Cell, macrophage, dendritic cell) by immunohistochemistry assay (CD3, CD4, CD8, CD20, CD16, CD56, granzyme B, cleaved caspase 3, and Ki-67) when distant tumor sample is obtained; if the sample volume is ample, additional immunohistochemistry assays will be performed for CD45RO, TIA-1, FoxP3, CD25, OX-40, CD57, CD1a, CD208, myeloperoxidase, CD68, COX-2, major histocompatibility complex (MHC) class I and MHC class II in Dr. Savitri Krishnamurthy's laboratory at MD Anderson.

OUTLINE:

Patients receive talimogene laherparepvec intratumorally (IT) on day 1. Cycles repeat every 3 weeks in cycle 1 and every 2 weeks thereafter in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of breast carcinoma
* Histological confirmation of recurrence of chest wall with or without distant metastasis disease
* Patients must have failed at least 1 systemic regimen or have clinical stable disease with capecitabine, hormonal therapy (with or without mTOR inhibitor or CDK4/6 inhibitor), or anti HER-2 therapy (trastuzumab, pertuzumab, ado-trastuzumab emtansine, lapatinib) for at least 2 months after their diagnosis of locoregional/metastatic disease
* Concurrent radiation therapy is permitted after the study treatment is initiated so long as the planned radiation field doesn't overlap with planned injection sites
* Eastern cooperative oncology group performance status (ECOG PS) 0-1
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L; if patient is taking CDK4/6 inhibitor or capecitabine, there is a need for maintaining ANC >= 1.0 consistently for at least 2 months without dose changes
* Platelet count >= 75 x 10^9/L, if patient is taking CDK4/6 inhibitor, ado-trastuzumab emtansine or capecitabine, there is a need for maintaining platelet count >= 75 x 10^9/L without dose changes
* Hemoglobin >= 8.0 g/L
* International normalization ratio (INR) or prothrombin time (PT) 1.5 x upper limit of normal (ULN), unless the subject is receiving anticoagulant therapy, in which case PT and partial thromboplastin time (PTT)/ activated PTT (aPTT) must be within therapeutic range of intended use of anticoagulants
* Serum creatinine =< 1.5 x upper limit of normal (ULN), OR 24-hour creatinine clearance >= 60 mL/min for subject with creatinine levels > 1.5 x ULN; (Note: creatinine clearance need not be determined if the baseline serum creatinine is =< 1.5 x ULN; creatinine clearance should be determined per institutional standard)
* Aspartate aminotransferase (AST) =< 2.5 x ULN if liver metastases present
* Alanine aminotransferase (ALT) =< 2.5 x ULN if liver metastases present
* Total bilirubin =< 1.5 x ULN, OR direct bilirubin =< ULN for a subject with total bilirubin level > 1.5 x ULN
* Subjects must be candidate for intralesional injection into cutaneous, subcutaneous or nodal tumors with or without image ultrasound guidance defined as one or more of the following at least 1 injectable lesion >= 5 mm in longest diameter, multiple injectable lesions that in aggregate have a longest diameter of >= 5 mm
* Female patients of childbearing potential must have negative urine pregnancy test no more than 3 days prior to starting study treatment
* Patients must be able and willing to give written informed consent

Exclusion Criteria:

* Patients who have operable disease with curable intent, and/or are candidates for radiation therapy for local control
* Patients receiving concurrent anti-cancer therapy (chemotherapy except capecitabine or ado-trastuzumab emtansine, immunotherapy) while taking study medication, or have previously received talimogene laherparepvec or any other oncolytic virus
* Patients with metastatic sites that requires chemotherapy (except capecitabine or ado-trastuzumab emtansine)
* Known active central nervous metastases; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids > 10 mg/day pf prednisone or equivalent; the exception does not include carcinomatosis meningitis which is excluded regardless of clinical stability
* More than three lesions per organ for visceral metastases except for lung or lymph node sites
* History or evidence of active autoimmune disease that has required systemic treatment (i.e., use of corticosteroids, immunosuppressive drugs or disease modifying agents); replacement therapy (eg, thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment for autoimmune disease
* Patients with concurrent disease or condition that would make them inappropriate for study participation, or any serious medical disorder that would interfere with patients' safety
* History of other malignancy within the past 5 years with the following exceptions: a) Adequately treated non melanoma skin cancer without evidence of disease at the time of enrollment b). Adequately treated cervical carcinoma in situ without evidence of disease at the time of enrollment c). Adequately treated breast ductal carcinoma in situ without evidence of disease at the time of enrollment d). Prostatic intraepithelial neoplasia without evidence of prostate cancer at the time of enrollment
* Patients with active infection and requiring intravenous (IV) or oral antibiotics
* Evidence of immune suppression as following:

  * Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)
  * Known leukemia or lymphoma
  * Primary immunodeficiency state such as severe combined immunodeficiency disease
  * Concurrent opportunistic infection
  * Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 7 days prior to the initiation of study treatment
  * Known hepatitis B or C infection
  * Congenital or acquired cellular and/or humoral immune deficiency
  * Other signs or symptoms of immune system suppression
* Active herpetic skin lesions or prior complication of herpes simplex virus (HSV)-1 infections (e.g. herpetic encephalitis or keratitis)
* Currently pregnant or breast-feeding, or planning to become pregnant during study treatment and through 3 months after the last dose of study treatment
* Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 3 months after the last dose of talimogene laherparepvec; (women of not childbearing potential: post-menopausal [age > 55 years with cessation of menses > 12 months or < 55 years but not spontaneous menses for at least 2 years or < 55 years and spontaneous menses within the past 1 year, but currently amenorrheic (eg, spontaneous or secondary to hysterectomy), and with postmenopausal gonadotropin levels (luteinizing hormone and follicle-stimulating hormone levels > 40 IU/L) or postmenopausal estradiol levels (< 5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved] or who have had a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy)
* Sexually active subjects and their partners unwilling to use male or female latex condom to avoid potential viral transmission during sexual contact while on treatment and within 30 days after treatment with talimogene laherparepvec
* Currently enrolled in another clinical trial for investigational drugs, procedures or device (excluding non-cancer treatment trials) or receipt of an investigational agent or device within 4 weeks of the initiation of study treatment
* Requires intermittent or chronic treatment with antiherpetic drugs, except for topical agents
* Patients who are known sensitive to any of the products or components to be administered during treatment with talimogene laherparepvec
* Chronic oral or systemic steroid medication use at a dose of > 10 mg/d of prednisone or equivalent (steroids with low systemic absorption [e.g. triamcinolone hexacetonide] injected into joint space are allowed)
* Prior therapy with tumor vaccine, or received live vaccine within 28 days prior to the initiation of study treatment
* Subjects who are unwilling to minimize exposure with his/her blood or other body fluids to individuals who are at higher risks for HSV-1 induced complications such as immunosuppressed individuals, individuals known to have HIV infection, pregnant women, or infants under the age of 3 months, during talimogene laherparepvec treatment and through 30 days after the last dose of talimogene laherparepvec
* Prior immunosuppressive, chemotherapy, radiotherapy (in which the field encompassed a planned injection site), biological cancer therapy (monoclonal antibodies), or major surgery within 28 days prior to enrollment or has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) grade 1 or better from adverse event due to cancer therapy administered more than 28 days prior to enrollment
* Prior radiotherapy in which the field does not overlap the injection sites or non-immunosuppressive targeted therapy within 14 days prior to enrollment or has not recovered to CTCAE grade 1 or better from adverse event due to cancer therapy administered more than 14 days prior to enrollment
* Patients who have extensive skin disease, defined as total area of skin involvement/ lesions that comprise > 10% of body surface area; skin involvement comprising > 5% to upper anterior chest wall or > 5% to upper posterior back is excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoto T Ueno, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 participants registered, 1 participant registered twice and 1 participant withdrew consent before initiating treatment to pursue alternate treatment.
Groups:
- Treatment (Talimogene Laherparepvec): Patients receive talimogene laherparepvec IT on day 1. Cycles repeat every 3 weeks in cycle 1 and every 2 weeks a total of at least 10 cycles, thereafter in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Talimogene Laherparepvec: Given IT
Period: Overall Study
Arm/Group | Treatment (Talimogene Laherparepvec)
Started | 9
Completed | 0
Not Completed | 9
Not completed — Disease Progression | 7
Not completed — Unrelated to study treatment | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 49 [39 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
Herpes Simplex Virus Type 1- HSV-1 Serology [Count of Participants; unit: Participants]
  Positive | 6
  Negative | 3
Type of breast cancer [Count of Participants; unit: Participants]
  Inflammatory Breast Cancer | 0
  Non-Inflammatory Breast Cancer | 9
Estrogen Receptor Status [Count of Participants; unit: Participants]
  Positive | 2
  Negative | 7
Progesterone Receptor Status [Count of Participants; unit: Participants]
  Positive | 2
  Negative | 7
HER2 Status [Count of Participants; unit: Participants]
  Positive | 1
  Negative | 8
Distant Metastases [Count of Participants; unit: Participants]
  No | 6
  Yes | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response Rate (ORR)
Description: Overall Response Rate defined as the rate of patients who achieved a partial response or complete response as the best response for the measurable and nonmeasurable disease. Evaluated using RECIST ver.1.1. Complete Response (CR): Disappearance of all target and non-target lesions at a minimum of 4 weeks. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter of the target lesions at a minimum of 4 weeks, taking as a reference the baseline sum of the longest diameter with target.
Time Frame: at the end of cycle 4 , cycle 8, and cycle 10, up to 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 9
Participants
  Complete Response | 0
  Partial Response | 0

2. Secondary Outcome: Median Progression-Free Survival
Description: Progressive disease is measured based on Response Evaluation Criteria (RECIST v1.1) beyond 10 cycles. Uncontrolled disease progression is defined as rapid growth of multiple measurable or non-measurable new lesions or sum of the longest diameter of existing targeted lesions is >40% from the baseline.
Time Frame: Time from treatment initiation until disease progression, uncontrolled disease progression or death. Maximum PFS follow-up for this study cohort was 3.9 months.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 9
days | 77 [63 to NA] — the upper bound of the Kaplan-Meier curve has not reached 50% yet therefore the upper bound of the median survival time cannot be estimated.

3. Secondary Outcome: Median Overall Survival
Description: Overall survival is defined as the time from treatment initiation until death. Estimated using the Kaplan-Meier method with 95% confidence intervals (CIs).
Time Frame: From the date of treatment initiation until 1 year after removal from the study or until death, whichever occurs first
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 9
days | 361 [240 to NA] — the upper bound of the Kaplan-Meier curve has not reached 50%yet therefore the upper bound of the median survival time cannot be estimated.

4. Secondary Outcome: Number of Adverse Events
Description: The number of Grade 2 or higher adverse events possibly, probably, or definitely related to T-VEC. Evaluated according to Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: before each cycle and 30 days after the last dose of trial treatment or before the initiation of a new anti-cancer treatment, whichever comes first
Measure: Number; unit: adverse events
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 9
adverse events
  Grade 2 | 29
  Grade 3 | 4

ADVERSE EVENTS:
Time Frame: From the date of treatment initiation until 30 days after the last dose of drug; All-Cause Mortality: From the date of treatment initiation until 1 year after removal from the study or until death, whichever occurs first.
Description: Grade 2 or higher non-hematologic AEs and grade 3 or higher hematologic AEs will be recorded upon observation by the investigator or reported by the patient (regardless of whether they are attributed to investigational product), documented in the patient's medical record, and recorded in CORe. Grade 2 or higher abnormal lab values will be recorded as AEs; and grade 1 abnormal laboratory values will not be recorded as AEs.
Arm/Group | Treatment (Talimogene Laherparepvec)
All-Cause Mortality (participants affected / at risk) | 6/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Talimogene Laherparepvec) (N=9)
Injection Site Infections (General disorders) | 2
Fever (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Talimogene Laherparepvec) (N=9)
Fatigue (General disorders) | 4
Fever (General disorders) | 2
Injection site reaction (General disorders) | 7
Tumor/injection site pain (General disorders) | 5
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Tumor/injection site infection (Gastrointestinal disorders) | 3
Myalgia (Gastrointestinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Lymphedema (Vascular disorders) | 3
Neutrophil count decreased (Investigations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT02658812/Prot_SAP_000.pdf